CLINICAL TRIAL: NCT04832048
Title: Comparative Clinical Trial on the Modifications of Cardiovascular Risk Factors When Performing Different Therapeutic Physical Exercise Programs With Different Intensities in Hypertensive and Dyslipidemic Patients.
Brief Title: Modifications in Cardiovascular Risk Factors When Performing Physical Exercise in Hypertensive and Dyslipidemic Patients
Acronym: ACTIVA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Católica San Antonio de Murcia (Other)
Responsible Party: Principal Investigator, Francisco Javier López Román, Principal Investigator, Universidad Católica San Antonio de Murcia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UCAMCFE-00021
Record Dates: First submitted 2021-03-31; First posted 2021-04-05 (Actual); Last update posted 2021-04-05 (Actual); Status verified 2016-09

CONDITIONS: Hypertension
Keywords: Blood Pressure monitoring; Primary care; Physical exercises; Training intensity
MeSH Terms: conditions — Hypertension; Motor Activity

STUDY DESIGN:
Intervention Model Description: A single-center, randomized, parallel-group, controlled, and open-label study was conducted.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High intensity training (HIT) group (Experimental): The HIT group performed the exercises with loads at 80-90% of HRF.
  Interventions: Other: Therapeutic physical exercise
- Low-moderate intensity training (LMIT) group (Experimental): The HIT group performed the exercises with the loads at 50-70% of the HRF
  Interventions: Other: Therapeutic physical exercise
- No training group (Placebo Comparator): They did not perform any type of programmed physical exercise during the study.
  Interventions: Other: No physical exercise

INTERVENTIONS:
Other: Therapeutic physical exercise — The physical training program was carried out 3 days a week in 1-hour sessions focused on basic endurance exercises (global body activities), strength (specific muscle region activities) and flexibility.
  Intensity was be determined by Maximum Heart Rate (HRF).
  Arms: High intensity training (HIT) group; Low-moderate intensity training (LMIT) group
Other: No physical exercise — No programmed physical exercise
  Arms: No training group

SUMMARY:
Single-center, randomized, parallel-group, controlled, open-label study. The aim of the study was to evaluate the effects of an exercise training program intervention of different intensities (high intensity versus low-moderate intensity) on blood pressure reduction as a complementary strategy in hypertensive individuals being treated with at least one antihypertensive drug.

DETAILED DESCRIPTION:
All participants included in the study were referred by their primary care physicians, who prescribed physical exercise as a healthy lifestyle intervention added to the antihypertensive regimens in the framework of the "ACTIVA-Murcia Program".

Participants in the HIT and LMIT groups followed the same physical training program, with the only difference being the intensity of the training. The program included two phases of physical exercise lasting 12 weeks and 16 weeks, respectively, separated by a 7-week rest period, which coincided with a holiday period. The times of both phases were not equal in terms of duration, since it is a community physical exercise program established by the Region of Murcia, and does not depend on the researchers.

The program was developed by graduates in Physical Activity and Sport Sciences, who were in charge of teaching the exercises and supervised each training session.

Participants assigned to the HIT and LMIT groups were given guidelines to continue physical exercise during the 7-week rest period, while participants in the control group were offered to participate in the program after the study.

ELIGIBILITY:
Inclusion Criteria:

* Age between 40 and 65 years.
* Under treatment with at least one antihypertensive drug for hypertension. Treatment should have lasted at least 12 months prior to inclusion in the study.
* Diagnosed with dyslipidemia under pharmacological treatment or with a specific hypercholesterolemia (> 200 mg/dL) in the past and a cholesterol level at the start of the study greater than 200 mg/dL.
* Patient in Primary Prevention.
* Subjects who do not develop physical exercise scheduled on a weekly basis.
* Subjects who have given written informed consent to participate in the study.

Exclusion Criteria:

* Serious or terminal illnesses.
* Diagnosis of ischemic and/or cerebrovascular heart disease.
* Presence of chronic diseases that prevent the performance of a physical exercise program or a stress test (disabling arthropathies, chronic moderate/severe pneumopathies, arrhythmias, etc).
* Severe mental illnesses: psychosis, severe depressive disorder, neurosis.
* Diabetes mellitus.
* Presence of absolute or relative contraindications dictated by the American College of Sports Medicine (ACSM, 1995), during the performance of the stress tests.
* Pregnant or breast-feeding women
* Inability to understand the informed consent.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2016-09-20 (Actual); Primary Completion 2017-06-12 (Actual); Study Completion 2019-12-20 (Actual)

PRIMARY OUTCOMES:
Ambulatory blood pressure monitoring | Measurements will be taken at baseline and 12 weeks (phase 1) and at baseline and 16 weeks (phase 2)
  Blood pressure is measured with a holter

SECONDARY OUTCOMES:
Systolic blood pressure | Measurements will be taken at baseline and 12 weeks (phase 1) and at baseline and 16 weeks (phase 2)
  Blood pressure is measured with a holter
Diastolic blood pressure | Measurements will be taken at baseline and 12 weeks (phase 1) and at baseline and 16 weeks (phase 2)
  Blood pressure is measured with a holter
Mean blood pressure | Measurements will be taken at baseline and 12 weeks (phase 1) and at baseline and 16 weeks (phase 2)
  Blood pressure is measured with a holter
Pulse pressure | Measurements will be taken at baseline and 12 weeks (phase 1) and at baseline and 16 weeks (phase 2)
  Blood pressure is measured with a holter
Lipid profile | Measurements will be taken at baseline and 12 weeks (phase 1) and at baseline and 16 weeks (phase 2)
  Blood samples
Antihypertensive medication | Measurements will be taken at baseline and 12 weeks (phase 1) and at baseline and 16 weeks (phase 2)
  Record of medication and dosage
Lipid lowering medication | Measurements will be taken at baseline and 12 weeks (phase 1) and at baseline and 16 weeks (phase 2)
  Record of medication and dosage
Control of dietary intake | A nutritional registry will be carried out. The nutritional intake of three days in two periods will be collected. One record at the beginning and another at the end, that is, six days.
  Diet source
Muscle function | Measurements will be taken at baseline and 12 weeks (phase 1) and at baseline and 16 weeks (phase 2)
  Isokinetic dynamometry.
Balance | Measurements will be taken at baseline and 12 weeks (phase 1) and at baseline and 16 weeks (phase 2)
  Force platform Kistler
Aerobic function | Measurements will be taken at baseline and 12 weeks (phase 1) and at baseline and 16 weeks (phase 2)
  Modified Balke-Ware protocol on a rolling mat
Framingham tables by category | Measurements will be taken at baseline and 12 weeks (phase 1) and at baseline and 16 weeks (phase 2)
  Physicians Global Assessment to measure cardiovascular risk

CONTACTS AND LOCATIONS:
Locations (1):
- Catholic University of Murcia, Murcia, Spain